CLINICAL TRIAL: NCT07386769
Title: Interpersonal Brain Function in Opioid Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Eric Garland, Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 813632
Record Dates: First submitted 2026-01-23; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: People Who Use Opioids/People With Opioid Use Disorder (OUD)
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation (Experimental): 20 minutes of guided meditation during the laboratory session involving mindfulness of breathing and lovingkindness practice.
  Interventions: Behavioral: Meditation
- Psychoeducation (Active Comparator): Psychoeducation about opioid neuropharmacology.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Meditation — 20 minutes of guided meditation during the laboratory session involving mindfulness of breathing and lovingkindness practice.
  Arms: Meditation
Behavioral: Psychoeducation — 20 minute psychoeducational script on the impact of opioid use on the brain.
  Arms: Psychoeducation

SUMMARY:
The purpose of this study is to assess dyadic physiological coherence and subjective empathic attunement during meditation practices and their association with opioid-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Persons, aged 18 or older
2. Current near daily use of prescribed or illicit opioid agonists or mixed opioid agonist-antagonists for ≥90 days
3. Must be able to speak and understand English

Exclusion Criteria:

1. Cognitive Impairment that would preclude participation in the research protocol
2. Active suicidal intent or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological synchrony | During the intervention and for 5 minutes afterwards
  Dyadic Neural Synchrony (DNS) across electrodes and dyads will be computed from EEG oscillations using established inter-brain connectivity metrics. DNS will be quantified as a dyadic coupling parameter computed from time-series features extracted from each participant's EEG activity. Higher DNS values indicate greater therapist-patient neural attunement.

SECONDARY OUTCOMES:
Interpersonal Attunement | During Intervention
  Interpersonal attunement measured by the Interpersonal Attunement Rating Scale, a 0-10 numeric rating scale to assess sense of connection with the other person (0=no attunement, 10=very high attunement).
Opioid Craving | Pre-Intervention, during Intervention, immediately post-Intervention, and at 1 month follow-up
  Opioid craving measured by 0-10 numeric rating scale (0=no craving, 10=extreme craving).
Opioid Use | Pre-Intervention, and 1 month Follow-Up
  Days of opioid use measured by the Timeline Followback Interview and completion of a urine drug toxicology screen.
Severity of Pain | Pre-Intervention, during Intervention, immediately post-Intervention, and at 1 month follow-up
  Pain rating measured by scores on Brief Pain Inventory, with higher scores indicating higher pain severity (min 0, max 10)
Affect | Pre-Intervention, during Intervention, and immediately post-Intervention.
  Positive and negative affect measured on a 0-10 numeric rating scale (0=low affect, 10=very high affect).
State Self-Transcendence | Pre-Intervention, during Intervention, immediately post-Intervention.
  Nondual awareness measured by the Nondual Awareness Dimensional Assessment Measure- State (NADA-S), with scores ranging from 0 to 30, with higher scores indicating greater self-transcendence
Metacognitive processes | Pre-Intervention, during Intervention, and immediately post-Intervention.
  Metacognitive Processes of Decentering Scale (MPODS), a 3-Item scale with scores ranging from 0 to 30, with higher scores indicating greater capacity for meta-awareness, non-reactivity, and disidentification.
Cardiac-autonomic synchrony | During the intervention and for 5 minutes afterwards
  Cardiac-autonomic synchrony (CAS) will be computed from heart rate variability. CAS will be quantified as a dyadic coupling parameter computed from time-series features extracted from each participant's R-R intervals. Higher CAS values indicate greater therapist-patient autonomic attunement.
Facial expression synchrony | During the intervention and for 5 minutes afterwards
  Facial Expression Synchrony (FES) will be assessed using automated facial expression analysis derived from computer-vision-based facial landmark and action-unit detection. FES will be quantified as a dyadic coupling parameter computed from time-series features extracted from each participant's facial expressions. Higher FES values indicate greater therapist-patient affective attunement

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garland, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will adhere to the NIH Grants Policy on Availability of Research Results: Publications, Intellectual Property Rights, and Sharing Biomedical Research Resources.
Time Frame: Data will become available after the publication of the main study findings from the final data set. Data will be made permanently available.
Access Criteria: Data will be made available upon reasonable request with a signed data access agreement.